CLINICAL TRIAL: NCT02140593
Title: Muscle Relaxation During Open Upper Abdominal Surgery - Can the Surgical Conditions be Optimized?
Brief Title: The Laparotomy Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Matias Vested Madsen, MD, research assistant, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lap2014NMB; 2014-001155-22 (EudraCT Number)
Record Dates: First submitted 2014-05-13; First posted 2014-05-16 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard neuromuscular blockade (Placebo Comparator): Rocuronium 0.6 mg/kg followed by bolus rocuronium according to standard treatment decided by the attending anesthetist combined with saline infusion (placebo).
  Interventions: Drug: Group STANDARD: Rocuronium 0.6 mg/kg followed by bolus rocuronium according to standard treatment combined with saline infusion (placebo).
- Deep neuromuscular blockade (Active Comparator): Rocuronium 0.6 mg/kg followed by rocuronium infusion with target level post tetanic count (PTC) of 0-1 combined with bolus saline (placebo) mimicking standard treatment.
  Interventions: Drug: Group DEEP: Rocuronium 0.6 mg/kg followed by rocuronium infusion with target level PTC 0-1 combined with bolus saline (placebo) mimicking standard treatment.

INTERVENTIONS:
Drug: Group STANDARD: Rocuronium 0.6 mg/kg followed by bolus rocuronium according to standard treatment combined with saline infusion (placebo).
  Arms: Standard neuromuscular blockade
Drug: Group DEEP: Rocuronium 0.6 mg/kg followed by rocuronium infusion with target level PTC 0-1 combined with bolus saline (placebo) mimicking standard treatment.
  Arms: Deep neuromuscular blockade

SUMMARY:
The depth of neuromuscular blockade (NMB) during surgery may cause a clinical dilemma between optimal surgical conditions and the risk of postoperative residual blockade.

The aim of the study is to investigate if intense NMB improves surgical conditions during operation in patients scheduled for elective open upper abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Elective open upper abdominal surgery
* Can read and understand Danish
* Informed consent

Exclusion Criteria:

* Known allergy to rocuronium or sugammadex
* Severe renal disease, defined by S-creatinine> 0.200 mmol/L, GFR < 30ml/min or hemodialysis
* Neuromuscular disease that may interfere with neuromuscular data
* Abdominal mesh with size larger than 5*5 cm
* Lactating or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matias V Madsen, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Aarhus University Hospital Nørrebrogade, Aarhus, Denmark

REFERENCES:
- [Derived] Madsen MV, Scheppan S, Mork E, Kissmeyer P, Rosenberg J, Gatke MR. Influence of deep neuromuscular block on the surgeons assessment of surgical conditions during laparotomy: a randomized controlled double blinded trial with rocuronium and sugammadex. Br J Anaesth. 2017 Sep 1;119(3):435-442. doi: 10.1093/bja/aex241. PMID 28969327
- [Derived] Madsen MV, Scheppan S, Kissmeyer P, Mork E, Rosenberg J, Gatke MR. Neuromuscular blockade for improvement of surgical conditions during laparotomy: protocol for a randomised study. Dan Med J. 2015 Oct;62(10):A5139. PMID 26441396

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Neuromuscular Blockade: Rocuronium 0.6 mg/kg followed by bolus rocuronium according to standard treatment decided by the attending anesthetist combined with saline infusion (placebo).
  Group STANDARD: Rocuronium 0.6 mg/kg followed by bolus rocuronium according to standard treatment combined with saline infusion (placebo).
- Deep Neuromuscular Blockade: Rocuronium 0.6 mg/kg followed by rocuronium infusion with target level post tetanic count (PTC) of 0-1 combined with bolus saline (placebo) mimicking standard treatment.
  Group DEEP: Rocuronium 0.6 mg/kg followed by rocuronium infusion with target level PTC 0-1 combined with bolus saline (placebo) mimicking standard treatment.
Period: Overall Study
Arm/Group | Standard Neuromuscular Blockade | Deep Neuromuscular Blockade
Started | 63 | 65
Completed | 63 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Neuromuscular Blockade | Deep Neuromuscular Blockade | Total
Number analyzed (Participants) | 63 | 65 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10) | 63 (11) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 34 | 38 | 72
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — body mass index (kg/m^2)
  kg/m^2 | 25 (5) | 26 (5) | 25 (5)
Previous abdominal surgery [Count of Participants; unit: Participants] | 39 | 46 | 85

OUTCOME MEASURES:

1. Primary Outcome: Surgical Rating Score
Description: The final score for the surgical conditions of a patient defined as the average of all scores provided during the surgical procedure. (Rated on a 5 point subjective rating scale; 1: extremely poor, 2: poor, 3: acceptable, 4: good, 5: optimal)
Time Frame: After randomization every 30 minutes during the operation from first incision to last suture of fascial closure, up to 300 minutes
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Standard Neuromuscular Blockade | Deep Neuromuscular Blockade
Number analyzed (Participants) | 63 | 65
units on a scale | 4 [1 to 5] | 4.75 [3 to 5]
Statistical Analysis 1: Comparison: Standard Neuromuscular Blockade vs Deep Neuromuscular Blockade; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.75

2. Secondary Outcome: The Surgical Rating Score During Fascial Closure
Description: After last suture of fascial closure surgical conditions are rated on a 5 point scale
Time Frame: Immediatly after fascial closure
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Standard Neuromuscular Blockade | Deep Neuromuscular Blockade
Number analyzed (Participants) | 63 | 65
units on a scale | 4 [1 to 5] | 5 [3 to 5]
Statistical Analysis 1: Comparison: Standard Neuromuscular Blockade vs Deep Neuromuscular Blockade; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 1.0

ADVERSE EVENTS:
Time Frame: Data collected from inclusion until 28 days after surgery by reviewing patient charts
Arm/Group | Standard Neuromuscular Blockade | Deep Neuromuscular Blockade
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/65
Other Adverse Events (participants affected / at risk) | 0/63 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes